CLINICAL TRIAL: NCT03662087
Title: Hypomethylating Agents + Donor Lymphocyte Infusion vs Donor Lymphocyte Infusion Preemptive Therapy Based on Minimal Residual Disease for Acute Leukemia Undergoing Allogenetic Hematopoietic Stem Cell Transplantation
Brief Title: HMA+DLI vs DLI Preemptive Therapy Based on MRD for AL Undergoing Allo-HSCT
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Principal Investigator, Qifa Liu, Prof., Nanfang Hospital, Southern Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HMA+DLI vs DLI-MRD-AL-2018
Record Dates: First submitted 2018-09-05; First posted 2018-09-07 (Actual); Last update posted 2018-09-07 (Actual); Status verified 2018-07

CONDITIONS: Minimal Residual Disease,Acute Leukemia, Hypomethylating Agents, Donor Lymphocyte Infusion, Allogeneic Hematopoietic Cell Transplantation
MeSH Terms: conditions — Neoplasm, Residual

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HMA+DLI (Experimental): For AL patients who achieved CR at pre-transplantation undergoing allo-HSCT, DLI was not given and immunosuppressant were withdrawn if patients were MRD persistently negative. MRD status were monitored every 30 days. If patients were MRD negative by Day+30 post-transplantation, MRD status would be continued to be monitored by Day+60. If patients were MRD positive by Day+30 post-transplantation, immunosuppressant were withdrawn. If MRD were persistently positive until Day+60 or MRD changed from negative by Day+30 to positive by Day +60 post-transplantation, HMA and DLI were given. DLI was given 48 hours after administration of HMA. DLI was given monthly until GVHD occurred or MRD became negative or a total of four times. If MRD changed from positive by Day+30 to negative by Day+60 post-transplantation, MRD status would be continued to be monitored by Day+90 post-transplantation. If patients were MRD positive by Day+90 post-transplantation, HMA and DLI were given as shown above.
  Interventions: Combination Product: HMA+DLI
- DLI (Experimental): For AL patients who achieved CR at pre-transplantation undergoing allo-HSCT, DLI was not given and immunosuppressant were withdrawn if patients were MRD persistently negative. MRD status were monitored every 30 days. If patients were MRD negative by Day+30 post-transplantation, MRD status would be continued to be monitored by Day+60 post-transplantation. If patients were MRD positive by Day+30 post-transplantation, immunosuppressant were withdrawn. If MRD were persistently positive until Day+60 or MRD changed from negative by Day+30 to positive by Day+60 post-transplantation, DLI was given. DLI was given monthly until GVHD occurred or MRD became negative or a total of four times. If MRD changed from positive by Day+30 to negative by Day+60 post-transplantation, MRD status would be continued to be monitored by Day+90 post-transplantation. If patients were MRD positive by Day+90 post-transplantation, DLI was given as shown above.
  Interventions: Biological: DLI

INTERVENTIONS:
Combination Product: HMA+DLI — HMA: Decitabine was administered at 20mg/m2/day for five consecutive days or Ara-C was administered at 75mg/m2/day for seven consecutive days. DLI was administered at a median dose of 1.0 (range 0.7-1.4) ×10*8 mononuclear cells/kg.
  Arms: HMA+DLI
Biological: DLI — DLI was administered at a median dose of 1.0 (range 0.7-1.4) ×10*8 mononuclear cells/kg.
  Arms: DLI

SUMMARY:
Allogeneic hematopoietic cell transplantation (Allo-HSCT) is an effective therapy for acute leukemia, but relapse is the most common problem affecting long-term survivors of allo-HSCT. Therapy options for relapse include stopping immune suppression, re-induction of chemotherapy, donor lymphocyte infusion (DLI) or combination therapy. In this prospective randomized controlled study, the safety and efficacy of hypomethylating agents (HMA) + DLI and DLI preemptive therapy based on minimal residual disease in acute leukemia undergoing allo-HSCT are evaluated.

DETAILED DESCRIPTION:
Allogeneic hematopoietic cell transplantation (Allo-HSCT) is an effective therapy for acute leukemia, but relapse is the most common problem affecting long-term survivors of allo-HSCT. Therapy options for relapse include stopping immune suppression, re-induction of chemotherapy, donor lymphocyte infusion (DLI) or combination therapy. One method of solving relapse is to intervene before hematologic or pathologic relapse occurs based on minimal residual disease (MRD) . DLI is an effective post-transplantation therapy based on MRD for relapse. Whether combination of hypomethylating agents (HMA) and DLI could improve outcomes remains unclear. In this prospective randomized controlled study, the safety and efficacy of HMA+DLI and DLI preemptive therapy based on minimal residual disease in acute leukemia undergoing allo-HSCT are evaluated.

ELIGIBILITY:
Inclusion Criteria:

- A patient age of 14-65 years. AL patients who achieved CR at pre-transplantation undergoing allo-HSCT. Subjects (or their legally acceptable representatives) must have signed an informed consent document indicating that they understand the purpose of and procedures required for the study and are willing to participate in the study.

Exclusion Criteria:

* AL patients who were in NR at pre-transplantation undergoing allo-HSCT. Any abnormality in a vital sign (e.g., heart rate, respiratory rate, or blood pressure). Patients with any conditions not suitable for the trial (investigators' decision).

Ages: 14 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-10 (Estimated); Primary Completion 2021-10 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
Relapse | 2 years
  Relapse was defined by reappearance of blasts in the peripheral blood, recurrence of BM blasts >5%, or development of extramedullary disease infiltrates at any site

SECONDARY OUTCOMES:
Disease-free survival (DFS) | 2 years
  DFS was defined as the time from transplantation to relapse or death in remission
Overall survival (OS) | 2 years
  OS was defined as the time from transplantation to death from all causes
Transplant-related mortality (TRM) | 2 years
  TRM was defined as death from any cause except relapse
Incidence of acute GVHD | 100 days
  Acute GVHD was graded according to standard criteria
Incidence of chronic GVHD | 2 years
  Chronic GVHD was assessed in patients alive after day 100

CONTACTS AND LOCATIONS:
Overall Officials: Qifa Liu, Principal Investigator — Nanfang Hospital, Southern Medical University
Locations (1):
- Department of Hematology,Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Yan CH, Liu DH, Liu KY, Xu LP, Liu YR, Chen H, Han W, Wang Y, Qin YZ, Huang XJ. Risk stratification-directed donor lymphocyte infusion could reduce relapse of standard-risk acute leukemia patients after allogeneic hematopoietic stem cell transplantation. Blood. 2012 Apr 5;119(14):3256-62. doi: 10.1182/blood-2011-09-380386. Epub 2012 Feb 14. PMID 22337715